CLINICAL TRIAL: NCT05254470
Title: Customer Survey of Athletic Trainers Who Utilize SAM Ultrasound Device in Routine Care
Brief Title: Real-World Experience of Patients Treated for Musculoskeletal Injuries With SAM in Routine Care
Status: Completed | Type: Observational
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-02-2021
Record Dates: First submitted 2022-02-05; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Musculoskeletal Injury; Pain, Chronic; Pain, Acute; Sport Injury; Soft Tissue Injuries; Arm Injury; Back Pain; Tendon Injuries; Muscle Injury
Keywords: Continuous Ultrasound; Sustained Acoustic Medicine; Musculoskeletal Injuries; Low Intensity Contiguous Ultrasound; Pain; Soft Tissue Injury
MeSH Terms: conditions — Chronic Pain; Acute Pain; Soft Tissue Injuries; Arm Injuries; Back Pain; Tendon Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pre-Low Intensity Continuous Ultrasound Treatment: Routine care for pain alleviation, range of motion and ability to return to work with traditional therapies from rehabilitation.
- Post-Low Intensity Continuous Ultrasound Treatment: Routine care of pain alleviation, range of motion and ability to return to work after treatment with low-intensity continuous ultrasound (LICUS) in conjunction with traditional therapies.
  Interventions: Device: Continuous Ultrasound

INTERVENTIONS:
Device: Continuous Ultrasound — 3MHz, 0.132W/cm2, 1.3W for 4 hours day delivered by an acoustic device
  Groups: Post-Low Intensity Continuous Ultrasound Treatment

SUMMARY:
The purpose of this study is to evaluate continuous ultrasound treatment with diclofenac coupling patch during routine care of musculoskeletal injuries which failed conservative treatment to better understand clinical utilization of the treatment on types of injuries, how the treatment helps patients (pain, function and quality of life), and information on healthcare provider ordering the therapy and general workflow.

Low-intensity continuous ultrasound (LICUS) is a bio regenerative technology used when normal rehabilitation is insufficient, applied with a wearable device (SAM, Zetroz Systems LLC) for daily use. The treatment provides long-duration ultrasound for approximately four hours. The objective of this study is to examine the real-world outcome data on symptoms improvement and return to function using SAM during routine care.

DETAILED DESCRIPTION:
ZetrOZ's SAM Ultrasound Device is a portable and wearable medical device which, when applied to various areas of the body, applies Low Intensity Therapeutic Ultrasound to deep tissues. The SAM device is currently used by a broad range of Athletic Trainers (ATs) in the United States to assist in the rehabilitation of injured athletes.

The purpose of this this study is to examine the real-world outcome data on symptoms improvement and return to function using SAM during routine care. This includes understanding utilization of the treatment (how often and how much time), how the treatment helps patients (rehabilitation and recovery), and information on SAM treatment augmenting conservative therapies.

ELIGIBILITY:
Inclusion Criteria:

* Work-related musculoskeletal injuries with limited improvement under traditional therapies

Exclusion Criteria:

* Healthy participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with work and sport related musculoskeletal injuries
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NRS) (0-10) | 0 - 4 weeks
  Change in pain severity over the time of treatment, 0 being lowest, and 10 being the worst pain.

SECONDARY OUTCOMES:
Global Health Improvement Score (GROC) (-7 to +7) | 0 - 4 weeks
  Quality of health care improvement satisfaction from intervention compared to conservative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rod Walters, EdD, Study Director — Walters Sports Medicine Inc
Locations (1):
- Sport & Orthopaedic Physical Therapy, Fairfield, Connecticut, United States

REFERENCES:
- [Background] Draper DO, Wells A, Wilk K. Efficacy of Sustained Acoustic Medicine as an Add-on to Traditional Therapy in Treating Sport-related Injuries : Case Reports. Glob J Orthop Res. 2020;2(4):545. Epub 2020 Sep 21. PMID 33043316
- [Background] Langer MD, Lewis GK Jr. Sustained Acoustic Medicine: A Novel Long Duration Approach to Biomodulation Utilizing Low Intensity Therapeutic Ultrasound. Proc SPIE Int Soc Opt Eng. 2015 May;9467:94670I. doi: 10.1117/12.2178213. PMID 30078928
- [Background] Madzia A, Agrawal C, Jarit P, Petterson S, Plancher K, Ortiz R. Sustained Acoustic Medicine Combined with A Diclofenac Ultrasound Coupling Patch for the Rapid Symptomatic Relief of Knee Osteoarthritis: Multi-Site Clinical Efficacy Study. Open Orthop J. 2020;14:176-185. doi: 10.2174/1874325002014010176. Epub 2020 Dec 18. PMID 33408796
- [Background] Winkler SL, Urbisci AE, Best TM. Sustained acoustic medicine for the treatment of musculoskeletal injuries: a systematic review and meta-analysis. BMC Sports Sci Med Rehabil. 2021 Dec 18;13(1):159. doi: 10.1186/s13102-021-00383-0. PMID 34922606
- [Derived] Jarit P, Klyve D, Walters R. Long Duration Sonophoresis of Diclofenac to Augment Rehabilitation of Common Musculoskeletal Injuries. Glob J Orthop Res. 2023;4(2):584. Epub 2023 Jan 20. PMID 36865667